CLINICAL TRIAL: NCT03730922
Title: The DBCG RT Recon Trial: Delayed-immediate Versus Delayed Breast Reconstruction in Early Breast Cancer Patients Treated With Mastectomy and Adjuvant Loco-regional Radiation Therapy. A Multicenter Randomized and Single Arm Clinical Trial
Brief Title: Delayed-immediate Versus Delayed Breast Reconstruction in Breast Cancer Patients With Mastectomy and Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Principal Investigator, Tove Filtenborg Tvedskov, Consultant, DMSc, Phd, associated professor, Danish Breast Cancer Cooperative Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBCG RT Recon
Record Dates: First submitted 2018-10-02; First posted 2018-11-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Neoplasm Female; Complication of Radiation Therapy; Breast Implant; Complications
Keywords: Breast cancer; Reconstruction; Post mastectomy radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study started as a randomized trial but was november 2023 changed for a prospective single arm tieal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Delayed-immediate reconstruction (Experimental): Primary Surgery: Skin sparing mastectomy (nipple sparing if appropriate) and axillary surgery according to guidelines or protocol. Reconstruction with silicone implant or expander covered by pectoral muscle and mesh or matrix.
  Delayed reconstruction: Final reconstruction with any reconstructive procedure - being it autologous or implant-based (one- or two-stage, +/- acellular dermal matrix (ADM)) - is performed 6-12 months after completion of chemotherapy and PMRT. Any contralateral procedure is allowed when doing the delayed surgery, but not in relation to the initial cancer surgery.
  Interventions: Procedure: Delayed-immediate reconstruction
- B: Delayed reconstruction (Active Comparator): Primary surgery: Total mastectomy and axillary surgery according to guidelines or protocol.
  Delayed reconstruction: 6-12 months after completion of PMRT: final recon-struction with any reconstructive procedure - being it autologous or implant-based (one-or two-stage, +/- ADM). Any contralateral procedure is allowed at any time point after PMRT has been delivered This arm has been closed nov 2023
  Interventions: Procedure: Delayed reconstruction

INTERVENTIONS:
Procedure: Delayed-immediate reconstruction — Skin sparing mastectomy and reconstruction with silicone implant or expander covered by pectoral muscle and mesh or matrix. Final reconstruction with any reconstructive procedure 6-12 months after completion of chemotherapy and RT.
  Arms: A: Delayed-immediate reconstruction
Procedure: Delayed reconstruction — Total mastectomy and delayed reconstruction:with any reconstructive procedure 6-12 months after completion of PMRT
  Arms: B: Delayed reconstruction

SUMMARY:
In breast cancer patients treated by mastectomy and adjuvant post-mastectomy radiation therapy (PMRT) reconstruction is often delayed until 6 - 12 month after completion of chemotherapy and PMRT, due to high risk of complication. In this trial the safety of the delayed-immediate reconstruction method is tested, where a skin sparing mastectomy and reconstruction with silicone implant is performed at primary surgery to save the native skin for the final delayed reconstruction.

DETAILED DESCRIPTION:
An increasing proportion of breast cancer patients treated by mastectomy wish for a breast reconstruction. If post-mastectomy radiation therapy is recommended, the reconstruction is often delayed until 6 - 12 months after completion of chemotherapy and radiation therapy due to risk of complication that might delay adjuvant treatment. At this time the native skin over the removed breast cannot be used in the reconstruction, resulting in a suboptimal aesthetic outcome. In the delayed-immediate reconstruction method, a skin sparing mastectomy and reconstruction with implant is performed at primary surgery, to save the native skin under radiation therapy, thereby improving the chance for a good aesthetic outcome at the final delayed reconstruction. In this trial breast cancer patients treated by mastectomy and loco-regional radiation therapy is randomized to either delayed reconstruction or delayed-immediate reconstruction. The complication rate as well as morbidity, aesthetic outcome and psychological well-being after delayed-immediate reconstruction will be compared with delayed reconstruction

ELIGIBILITY:
Inclusion Criteria:

* Woman >18 years who are offered a mastectomy for invasive breast can-cer pT1-3, pN0-N3, M0 and wish reconstruction. The patient can be inclu-ded no matter the status of estrogen receptor, progesterone receptor, malignancy grade, and HER2 status.
* The patient is a candidate for loco-regional radiation therapy according to national or institutional guidelines.
* Highly selected patients with inflammatory breast cancer, namely those with complete or near complete response to neoadjuvant systemic thera-py judged by imaging and clinical examination before surgery. Any skin edema and clinical signs of skin involvement must have disappeared during systemic therapy. It is highly recommended that the decision to offer an inflammatory breast cancer patient inclusion in the DBCG RT Recon trial is made during a multidisciplinary team conference.
* Adjuvant systemic therapy with chemotherapy, endocrine therapy, anti-HER2 treatment and other targeted therapies used in the adjuvant setting either as new standard or as part of a trial during the course of the trial is accepted.
* Neoadjuvant chemotherapy and primary systemic therapy of an operable breast cancer is accepted.
* Patient with previous non-breast malignancy is accepted if the patient has been without disease minimum 5 years, and the treating oncologist esti-mates a low risk of recurrence. Patients with the following diseases can be accepted despite less than 5 years disease free interval: carcinoma in situ cervicis, carcinoma in situ coli, melanoma in situ, basal cell carcino-ma of the skin, squamous cell carcinoma of the skin.
* Life expectancy minimum 10 years.

Exclusion Criteria:

* Pregnant or lactating.
* Previous breast cancer or Ductal carcinoma in Situ (DCIS).
* Bilateral breast cancer.
* Previous radiation therapy to the chest region.
* Previous non-breast malignancy (not including carcinoma in situ of the cervix or colon, melanoma in situ, basal cell carcinoma of the skin, and squamous cell carcinoma of the skin) within 5 years.
* Conditions indicating that the patient cannot go through breast reconstruction, the radiation therapy or follow up.
* Not being able to participate due to language or other personal issues.
* Life expectancy less than 10 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 590 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complications with surgical intervention | 1 year after final reconstruction
  Number of patients with complication deeming surgical intervention necessary (excluding percutaneous drainage and antibiotic treatment for inflammation in cases without need for open drainage):
  * Infection
  * Hematoma
  * Loss of implant/expander
  * Necrosis
  * Seroma

SECONDARY OUTCOMES:
Number of patients with complications without surgical intervention | 1 year after final reconstruction
  Number of patients with complication (Infection with need for antibiotics and/or necrosis) without intervention necessary
Depression | 10 years post-final reconstruction
  Degree of Depression measured by Becks Depression Inventory, BDII using a scale from 1 to 4, 4 being the worst
Fear of cancer recurrence | 10 years post-final reconstruction
  Fear of cancer recurrence measured by Concerns About Recurrence Questionnaire-3 (CARQ-3 ) on a scale from 1 to 10, 10 worst (fear all the time)
Patient´s satisfaction and quality of life (QoL) | 10 years post-final reconstruction
  Patient satisfaction and QoL measures by the BREAST-Q-instruments on a scale from 1 to 5, 5 being worst
Timely initiation of adjuvant therapy | 1 year
  Time from primary surgery to start of adjuvant therapy
Degree of patient reported morbidity regarding body image, painsensory disturbanses and feeling og lymphoedema | 10 years post-final reconstruction
  Patient reported morbidity measured by a questionnaire. The prevalence of pain will be assessed on a 0-10 numerical rating scale (NRS) and reported as: 'light pain' NRS 1-3; 'moderate pain' NRS 4-6; and 'severe pain' NRS 7-10. Sensory disturbances will be assessed by a dichotomous 'yes/no' question,. Lymphoedema will be assessed on a 0-10 numerical rating scale, 10 being worst. Body image will be assessed on a 0-7 numerical rating scale, 7 being best.
Number of patients with lymphoedema | 10 years post-final reconstruction
  Difference in arm circumference between arms 15 cm/10 cm proximal/distal to the olecranon bilaterally. Any difference ≥10% defines lymhoedema.
Number of patients with restricted range of motion of the shoulder | 10 years post-final reconstruction
  Differences between arms in range of motion of the shoulder measured at abduction/flexion with the patient sitting in front of a poster with a circle with degrees 0-180˚.Any difference ≥10 degrees defines defines restricted motion
Number of patients with capsular contracture | 10 years post-final reconstruction
  Degree of capsular Contracture using Baker grading
Aesthetic outcome | 10 years post-final reconstruction
  Aesthetic outcome scored bt the physician using breast Photo, on a scale from 0 to 3, 3 being worst

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte V Offersen, Professor, Study Director — DBCG; Tove F Tvedskov, DMSc, Principal Investigator — DBCG; Tine Damsgaard, Professor, Study Director — DBCG; Peer Christiansen, Professor, Study Director — DBCG; Majbrit Jensen, MSc, Study Director — DBCG
Locations (8):
- Denmark (8):
  - Åbenrå Sygehus, Aabenraa
  - Ålborg Universitetshospital, Aalborg
  - Århus Universitets Hospital, Aarhus
  - Gentofte Hospital/Herlev Hospital, Copenhagen
  - Esbjerg Sygehus, Esbjerg
  - Sjællands Universitetshospital, Roskilde
  - Vejle Sygehus, Vejle
  - Viborg Sygehus, Viborg

REFERENCES:
- [Derived] Kaidar-Person O, Nissen HD, Yates ES, Andersen K, Boersma LJ, Boye K, Canter R, Costa E, Daniel S, Hol S, Jensen I, Lorenzen EL, Mjaaland I, Nielsen MEK, Poortmans P, Vikstrom J, Webb J, Offersen BV. Postmastectomy Radiation Therapy Planning After Immediate Implant-based Reconstruction Using the European Society for Radiotherapy and Oncology-Advisory Committee in Radiation Oncology Practice Consensus Guidelines for Target Volume Delineation. Clin Oncol (R Coll Radiol). 2021 Jan;33(1):20-29. doi: 10.1016/j.clon.2020.09.004. Epub 2020 Sep 26. PMID 32988717